CLINICAL TRIAL: NCT04435379
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multicentre, Clinical Trial to Assess the Efficacy and Safety of VPM1002 in Reducing Hospital Admissions and/or Severe Respiratory Infectious Diseases in Elderly in the SARS-CoV-2 Pandemic by Modulating the Immune System
Brief Title: Study to Assess VPM1002 in Reducing Hospital Admissions and/or Severe Respiratory Infectious Diseases in Elderly in COVID-19 Pandemic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Serum Life Science Europe GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VPM1002-DE-3.07CoV; 2020-001675-33 (EudraCT Number)
Record Dates: First submitted 2020-06-16; First posted 2020-06-17 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Infection, Respiratory Tract
Keywords: infectious respiratory diseases
MeSH Terms: conditions — Respiratory Tract Infections | interventions — VPM1002 recombinant BCG vaccine

STUDY DESIGN:
Intervention Model Description: Subjects who fulfil the inclusion/exclusion criteria will be centrally randomized in a 1:1 ratio to receive a single dose (0.1 ml) of either VPM1002 or Placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The reconstitution of trial intervention will be done by unblinded site personnel who will not be involved in the collection or evaluation of outcome data. Administration of the trial intervention will be done by blinded site personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VPM1002 (Experimental): The active ingredient of the recombinant BCG vaccine, VPM1002, is Mycobacterium bovis rBCGΔureC::hly, freeze-dried and standardized to the number of viable mycobacteria (colony forming units; CFU) per application.
  Dose: 2-8 x 10e5 CFU VPM1002 administered in 0.1 ml reconstituted suspension.
  Interventions: Biological: VPM1002
- Placebo (Placebo Comparator): Physiological saline 0.1ml
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VPM1002 — The investigational product will be administered via intradermal injection with a 1.0-ml syringe, sub-graduated into hundredths of ml (1/100 ml), and fitted with a short bevel needle (25G/0.50 mm or 26G/0.45 mm, 10 mm in length).
  Arms: VPM1002
Biological: Placebo — The investigational product will be administered via intradermal injection with a 1.0-ml syringe, sub-graduated into hundredths of ml (1/100 ml), and fitted with a short bevel needle (25G/0.50 mm or 26G/0.45 mm, 10 mm in length).
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate whether vaccination of elderly with VPM1002 could reduce hospital admissions and/or severe respiratory infectious diseases in the SARS-CoV-2 pandemic .

VPM1002 is a vaccine that is a further development of the old Bacillus Calmette-Guérin (BCG) vaccine, which has been used successfully as a vaccine against tuberculosis for about 100 years, especially in developing countries. VPM1002 has been shown in various clinical studies to be significantly safer than the BCG vaccine.

VPM1002 strengthens the body's immune defence and vaccination with BCG reduces the frequency of respiratory diseases. It is therefore assumed that a VPM1002 vaccination could also provide (partial) protection against COVID-19 disease caused by the "new corona virus" SARS-CoV 2.

DETAILED DESCRIPTION:
Based on the evidence that BCG [Bacille Calmette-Guérin] vaccine

1. can potentiate immune responses to other vaccines through induction of trained innate immunity and heterologous adaptive immunity, and
2. can reduce the incidence of respiratory infections, exert antiviral effects in experimental models, and reduce viremia in an experimental human model of viral infection, it is hypothesized that BCG vaccination may induce (partial) protection against the susceptibility to and/or severity of SARS-CoV-2 infections.

VPM1002 is being developed with the aim to replace BCG by a vaccine that has a better safety profile and superior efficacy. Evidence from pre-clinical and clinical studies demonstrate that VPM1002 is safer and is more immunogenic than the existing BCG vaccine (for more information, please revert to the IB). It is therefore anticipated that VPM1002 will also perform better in reducing the severity of the symptoms of an infection with the SARS-CoV-2 than the BCG vaccine. Further, manufacturing of VPM1002 using state-of-the-art production methods will help hasten the production of millions of doses in a very short time and thus would be beneficial in the current SARS-CoV-2 pandemic situation.

The current trial will assess the efficacy and safety of VPM1002 to reduce the hospital admissions and clinical consequences of SARS-CoV-2 infections in the elderly population in the SARS-CoV-2 pandemic by modulating the immune system.

A total of 2038 adults aged 60 or above will be enrolled across involved clinical trial sites in Germany. Informed consent will be obtained from the subjects willing to take part in the trial. This will be followed by assessment of the eligibility criteria. Subjects who fulfil the inclusion/exclusion criteria will be centrally randomized in a 1:1 ratio to receive a single dose (0.1 ml) of either VPM1002 or Placebo.

All subjects will be requested to sign into a web-based tool designed for this trial. Every subject is encouraged to name a designated caregiver who may provide follow-up data in case of hospitalisation or severe illness of the study subject. All subjects will be followed-up entirely remotely. The questionnaires will be designed to collect data regarding hospitalisation, adverse events (AE)/serious adverse events (SAE), ICU admissions and other secondary endpoints. The investigators will review the outcome and safety data.

The duration of follow-up will be 240 days. Subjects with confirmed SARS-CoV-2 infection (with or without symptoms) will be followed for at least 6 weeks (from the date of test result), independent of the total trial duration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult (≥ 60 years)
2. Subject is contractually capable, able to understand information on study and has signed informed consent sheet
3. Subject has access to an internet-enabled electronic device

Exclusion Criteria:

1. Known active or latent Mycobacterium tuberculosis infection
2. Fever (> 38 °C) or respiratory tract infection within the past 24 hours
3. Current active viral or bacterial infection
4. Expected vaccination during the study period; vaccinations against influenza and pneumococcal disease are allowed with ≥ 4 weeks between these vaccinations and the trial vaccination
5. Participation in another interventional study within 30 days before screening and during this study
6. Known hypersensitivity or allergy to (components of) the VPM1002 vaccine or serious adverse reactions to prior Bacille Calmette-Guérin (BCG) administration
7. Severely immunocompromised subjects, including:

   1. subjects with known infection by the human immunodeficiency virus (HIV-1);
   2. subjects with solid organ transplantation;
   3. subjects with bone marrow transplantation;
   4. subjects under chemotherapy, immunotherapy, or radiotherapy;
   5. subjects with primary immunodeficiency;
   6. treatment with any anti-cytokine therapies;
   7. treatment with oral or intravenous steroids defined as daily doses of 10 mg prednisone or equivalent for longer than 3 months, or likely use of oral or intravenous steroids in the next 4 weeks;
8. History of malignancies, unless the subject has been free of the disease for ≥ 2 years; exception: subjects with adequately treated basal or squamous cell cancer or other localized non-melanoma skin cancer and adequately treated carcinoma in situ of the cervix may participate in the trial
9. Previous positive SARS-CoV-2 test result
10. Person is an employee of the sponsor, a relative of the sponsor or investigator, or is employed in the same department as the investigator

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2038 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Number of days with severe respiratory disease at hospital and/or at home | From day 0 to day 240

SECONDARY OUTCOMES:
Cumulative incidence of hospital admissions | From day 0 to day 240
Cumulative incidence of documented SARS-CoV-2 infection | From day 0 to day 240
Number of days with self-reported fever (≥ 38 ºC) | From day 0 to day 240
Number of days with self-reported acute respiratory symptoms | From day 0 to day 240
Cumulative incidence of self-reported acute respiratory symptoms | From day 0 to day 240
Cumulative incidence of death for any reason | From day 0 to day 240
Cumulative incidence of death due to documented SARS-CoV-2 infection | From day 0 to day 240
Cumulative incidence of ICU admission for any reason | From day 0 to day 240
Cumulative incidence of ICU admission due to documented SARS-CoV-2 infection | From day 0 to day 240
Cumulative incidence of hospital admission due to documented SARSCoV- 2 infection | From day 0 to day 240

CONTACTS AND LOCATIONS:
Overall Officials: Leander Grode, Dr. rer. nat., Study Director — Serum Life Science Europe GmbH
Locations (12):
- Germany (12):
  - Hautarztpraxis Dres. Leitz & Kollegen, Stuttgart, Baden-Wurttemberg
  - MECS Cottbus GmbH, Cottbus, Brandenburg
  - Studienzentrum Dr. Keller, Frankfurt am Main, Hesse
  - Klinische Forschung Hannover Mitte GmbH, Hanover, Lower Saxony
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Medizentrum Essen Borbeck, Essen, North Rhine-Westphalia
  - BAG Dres. med. Quist PartG, Mainz, Rhineland-Palatinate
  - SIBAmed GmbH & Co. KG, Leipzig, Saxony
  - SocraTec R&D GmbH, Erfurt, Thuringia
  - emovis GmbH, Berlin
  - Klinische Forschung Berlin GbR, Berlin
  - Klinische Forschung Hamburg GmbH, Hamburg

IPD SHARING:
Plan to Share IPD: No
There is uncertainty whether the European Union General Data Protection Regulation allows dissemination of individual participant data to other researchers. Some reasons why the EU Regulation would not allow this are the lack of suitable safeguards when personal data are transferred to any researcher asking for it and the impairment of the rights of the subjects for erasure of their data once they are disseminated.

REFERENCES:
- [Derived] Blossey AM, Bruckner S, May M, Parzmair GP, Sharma H, Shaligram U, Grode L, Kaufmann SHE, Netea MG, Schindler C. VPM1002 as Prophylaxis Against Severe Respiratory Tract Infections Including Coronavirus Disease 2019 in the Elderly: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Multicenter Clinical Study. Clin Infect Dis. 2023 Apr 3;76(7):1304-1310. doi: 10.1093/cid/ciac881. PMID 36358012